CLINICAL TRIAL: NCT07077824
Title: Effect of Stellate Ganglion Block on Arterial Catheterization Complications in Selected Group of Patients Undergoing Elective Cardiac Surgeries
Acronym: stellate block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, abdallah mahmoud zaki soudi, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: fmasu R156/2025
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery
Keywords: stellate ganglion block; femoral radial gradient; arterial catheterization complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block group (Experimental): Patients will receive left stellate ganglion block US guided after induction of anesthesia and intubation and after insertion of Rt IJV CVL and before skin incision
  Interventions: Procedure: Stellate Ganglion Block Injection with Bupivicaine
- Control group (No Intervention): Patients will undergo the surgery according to practised protocol

INTERVENTIONS:
Procedure: Stellate Ganglion Block Injection with Bupivicaine — Patients will receive left stellate ganglion block US guided after induction of anesthesia and intubation and after insertion of Rt IJV CVL and before skin incision
  Arms: Stellate Ganglion Block group

SUMMARY:
Radial artery catheterization is the usual method for invasive monitoring in cardiac surgeries. Although it is relatively safe, complications do happen. Hematoma and ischemia are well known complications. Also, radial-to-femoral arterial pressure gradient (RFAPG) post bypass is a common event which affect management of a critical patient in a critical time. the study examines the effect of left stellate ganglion block (LSGB) on decreasing radial artery complications in cardiac surgeries

DETAILED DESCRIPTION:
Invasive blood monitoring is an essential prerequisite in all cardiac surgeries where the radial artery is the most common one used. It is easily accessible, apart from important nerves and has a well-known safe profile.

As perfection is an unattainable dream, radial artery complications do happen ranging from spasm, occlusion, hematoma formation and dissection Although incidence of ischemia post radial artery occlusion is not as common as the occlusion, serious effects do happen as reported digital necrosis and the need to do below elbow amputation in one case Patients undergoing cardiac surgeries usually suffers from many risk factors for Ischemic complications as risk of hypotension and use of vasoconstrictors The use of vasoconstrictors is more expected in patients with preoperative decreased Left Ventricle (LV) function (≤30%), moderate to severe Pulmonary Hypertension (PH), multiple procedures and prolonged bypass time.

Also, a complication that is relatively common in open heart surgeries is the central to radial artery pressure gradient that is usually encountered post bypass and may last for some time after and may affect up to 45% of patients in cardiac surgeries.

Usually the pressure gradient is for favor of the radial artery in awake patients due to the vascular resistance, but many theories tried to explain the cause of the opposed gradient post bypass. One theory related the issue to Vasoconstriction of the brachial artery.

Over the last few years, there were some studies, which investigated the effect of regional anesthesia techniques such as thoracic epidural anesthesia (TEA) and stellate ganglion block (SGB) for sympatholysis in cardiac surgeries The SGB with local anesthetics have been widely used to provide pain relief to treat vascular spastic disorders of upper limbs, chronic pain conditions and treatment of refractory angina The SGB has also been used for increasing radial artery (RA) blood flow and preventing RA spasm by sympathetic blockade in coronary artery bypass surgery In the current study, SGB will be studied regarding its effect in minimizing the occurrence of complications related to arterial catheterization in selected patients in cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

* • Multiple procedures with expected prolonged bypass time (>100 min)

  * EF< 35%
  * Moderate or severe Pulmonary hypertension

Exclusion Criteria:

* • Patient not willing to participate in the study.

  * History of strokes / Transient ischaemic attacks
  * History of Glaucoma.
  * History of allergy to local anaesthetic drugs.
  * Pre-existing contralateral phrenic nerve palsy.
  * Patients with existing coagulopathy.
  * BMI >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of arterial ischemia | from end of surgery till hospital discharge aproximately one week
  Incidence of arterial ischemia in form of colour changes and confirmed by arterial duplex

SECONDARY OUTCOMES:
• Incidence of radial to femoral artery pressure gradient | from weaning from cardiopulmonary bypass till transferal to icu aproximately 1-2 hours
  • Incidence of radial to femoral artery pressure gradient which is defined as one of the following: >25 mmhg in systolic BP or > 10 mmhg in mean BP that is sustained for > 5 minutes either before, on or after CPB

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt